CLINICAL TRIAL: NCT01972503
Title: A Prospective,Randomized Control Trial of Intraoperative Intraportal Chemotherapy (5-FU and Oxaliplatin) Combined With Adjuvant Chemotherapy to Prevent Liver Metastasis in Patients Receiving Curative Colorectal Cancer Resection.
Brief Title: Intraoperative Intraportal Chemotherapy Combined With Adjuvant Chemotherapy for Stage II and III Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Jianmin Xu, PhD Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Octree Study
Record Dates: First submitted 2013-09-23; First posted 2013-10-30 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms
Keywords: Colorectal Neoplasms; Liver; Neoplasm Metastasis; Tegafur; oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms | interventions — Fluorouracil; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Experimental): Patients with stage II or stage III colorectal cancer (CRC) were randomly assigned to two arms. In ARM A, patients accepted intraoperative intraportal infusion of 5-FU 1g and oxaliplatin 100mg + curative resection+mFOLFOX6.
  Interventions: Drug: 5-FU and oxaliplatin; Procedure: colorectal cancer resection+ adjuvant chemotherapy (mFOLFOX6)
- ARM B (Active Comparator): Patients with stage II or stage III colorectal cancer (CRC) were randomly assigned to two arms. In arm B, patients accepted curative resection + mFOLFOX6 alone.
  Interventions: Procedure: colorectal cancer resection+ adjuvant chemotherapy (mFOLFOX6)

INTERVENTIONS:
Drug: 5-FU and oxaliplatin — Patients with stage II or stage III colorectal cancer (CRC) were randomly assigned to two arms. In arm A, patients accepted intraoperative intraportal infusion of 5-FU 1g and oxaliplatin 100mg+ curative resection + mFOLFOX6.
  Arms: ARM A
Procedure: colorectal cancer resection+ adjuvant chemotherapy (mFOLFOX6) — Patients with stage II or stage III colorectal cancer (CRC) were randomly assigned to two arms. All patients in both arms accept curative resection of colorectal cancer,and accept standard adjuvant chemotherapy (mFOLFOX6).

SUMMARY:
In this study, the investigators assessed whether intraoperative Intraportal infusion of 5-FU and oxaliplatin is able to prevent liver metastasis in patients receiving curative colorectal cancer resection.

DETAILED DESCRIPTION:
In this study, the investigators assessed whether intraoperative Intraportal infusion of 5-FU and oxaliplatin is able to prevent liver metastasis and improve survival in patients with Stage II or Stage III colorectal cancer without apparent liver metastasis based on a thorough preoperative evaluation.

Patients with stage II or stage III colorectal cancer (CRC) were randomly assigned to two arms.Arm A: 5-FU 1g and oxaliplatin 100mg + curative resection (study group, n=132). Arm B: curative resection alone (control group, n=132).Follow-up: X-ray, US, CT, blood test, colonoscopy,every 3months.

The study endpoints were disease-free survival, overall survival, and liver metastasis-free survival as evaluated by intent-to-treat analysis.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 and ≤ 75 years and with histologically proven adenocarcinoma of the colon or rectum
2. WHO performance status of 0 or 1
3. Stage II (T3-4, N0, M0) or Stage III (T0-4, N1-2, M0) disease (according to the 1997 revision of the International Union Against Cancer TNM staging system) as determined by a preoperative evaluation that included colonoscopy and an abdominal computed tomography (CT) scan
4. Written informed consent for participation in the trial.

Exclusion criteria

1. has prior other malignant cancer
2. has severe major organ dysfunction
3. has prior cancer therapy before surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-06; Primary Completion 2013-09 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
3 years disease-free survival | 3 years after operation
  PFS will be defined as the period from the first day of CRC resection to the date of disease recurrence or to death.

SECONDARY OUTCOMES:
3 years overall survival and metastasis-free survival | 3 years after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chang W, Wei Y, Ren L, Zhong Y, Yu Y, Chen J, Zhu D, Ye L, Qin C, Zhao N, Niu W, Qin X, Xu J. Randomized Controlled Trial of Intraportal Chemotherapy Combined With Adjuvant Chemotherapy (mFOLFOX6) for Stage II and III Colon Cancer. Ann Surg. 2016 Mar;263(3):434-9. doi: 10.1097/SLA.0000000000001374. PMID 26465781